CLINICAL TRIAL: NCT04601688
Title: Study on Branch Retinal Vein Occlusion Patients Receiving Bevacizumab and Dexamethasone or Bevacizumab Only on Naive Eyes.
Brief Title: Branch Retinal Vein Occlusion (BRVO) Treatment With Bevacizumab and Dexamethasone or Bevacizumab Only.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: He Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ME-260620
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Branch Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — Bevacizumab; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BRVO: Bevacizumab and intravitreal Dexamethasone (Experimental): Participants with BRVO will receive a combination of Bevacizumab and intravitreal Dexamethasone.
  Interventions: Drug: Bevacizumab Ophthalmic and Intravitreal Dexamethasone
- BRVO: Bevacizumab (Active Comparator): Participants with BRVO will receive Bevacizumab only.
  Interventions: Drug: Bevacizumab Ophthalmic

INTERVENTIONS:
Drug: Bevacizumab Ophthalmic and Intravitreal Dexamethasone — Pro re nata patients with BRVO will initially receive Bevacizumab and intravitreal Dexamethasone. And then depending on their clinical status of BRVO, Bevacizumab will be injected.
  Other Names: Avastin®; Ozurdex®
  Arms: BRVO: Bevacizumab and intravitreal Dexamethasone
Drug: Bevacizumab Ophthalmic — Pro re nata patients with BRVO will receive Bevacizumab. And then depending on their clinical status of BRVO, Bevacizumab will be injected.
  Other Names: Avastin®
  Arms: BRVO: Bevacizumab

SUMMARY:
The aim of this study is to evaluate the visual outcome and prognostic factors after intraocular injections of Bevacizumab or combination of Bevacizumab And Dexamethasone under pro re nata treatment regimen for Branch Retinal Vein Occlusion (BRVO) patients.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the clinical outcome after intraocular injections of Bevacizumab or combination of Bevacizumab and Dexamethasone under pro re nata treatment regimen for the patients with Branch Retinal Vein Occlusion (BRVO) patients. Mean change of logarithm of the minimal angle of resolution (logMAR) visual acuity (VA), central foveal thickness (CFT), contrast sensitivity (CS) as well as predictive factors including best-corrected visual acuity (BCVA), vision related questionnaires and various other ocular parameters will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any study assessment is performed
2. Diagnosis of visual impairment exclusively due to ME secondary to BRVO
3. BCVA score at Screening and Baseline between 10/40 (0.5) to 20/400 (0.05) on the Snellen chart.
4. Central foveal thickness (CFT) ≥ 300 µm
5. Naive Eyes

Exclusion Criteria:

1. Pregnant or nursing (lactating) women
2. Stroke or myocardial infarction less than 3 months before Screening
3. Uncontrolled blood pressure defined as systolic value of >160 mm Hg or diastolic value of >100 mm Hg at Screening or Baseline.
4. Any active periocular or ocular infection or inflammation at Screening or Baseline in either eye
5. Uncontrolled glaucoma at Screening or Baseline or diagnosed within 6 months before Baseline in either eye
6. Neovascularization of the iris or neovascular glaucoma in the study eye
7. Use of any systemic or ocular antivascular endothelial growth factor (anti-VEGF) drugs within 6 months before Baseline
8. Panretinal laser photocoagulation performed, anticipated or scheduled in the study eye
9. Focal or grid laser photocoagulation in the study eye
10. Use of intra- or periocular corticosteroids (including sub-Tenon) or ocular anti-VEGF treatment within 3 months before Screening in the study eye
11. Any use of intraocular corticosteroid implants (eg, dexamethasone [Ozurdex®], fluocinolone acetonide [Iluvien®]) in the study eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-10-31 (Estimated); Primary Completion 2021-03-02 (Estimated); Study Completion 2021-09-17 (Estimated)

PRIMARY OUTCOMES:
Mean change in monocular BCVA in the treatment eye | Baseline, 1 week, 1month, 2 months, 3 months, and 6 months.
  Monocular BCVA in the treatment eye is assessed by using ETDRS visual acuity charts at 4 meters is assessed and compared.
Mean change in binocular BCVA | Baseline, 1 week, 1month, 2 months, 3 months, and 6 months.
  Binocular BCVA is assessed by using ETDRS visual acuity charts at 4 meters is assessed and compared.

SECONDARY OUTCOMES:
Mean change in central subfield retinal thickness | Baseline, 1 day, 1 week, 1month, 2 months, 3 months, and 6 months.
  Mean change in central subfield retinal thickness in the study eye, as determined by spectral domain optical coherence tomography (OCT) is assessed and compared.
Change in Humphrey 10-2 visual field in the treatment eye | Baseline, 1 day, 1 week, 1month, 2 months, 3 months, and 6 months.
  Mean deviation (MD) of the Humphrey 10-2 visual field is assessed by a Humphrey 10-2 visual field test and compared.
Number of Bevacizumab. Treatments | Day 1 through Month 6
  Number of injections provided to the patients during the 6 month period.
Mean change in NEI VFQ25 | Baseline, 1 day, 1 week, 1month, 2 months, 3 months, and 6 months.
  Scores from NEI VFQ25 questionnaire is assessed and compared.
Mean change in EQ-5D 5L | Baseline, 1 day, 1 week, 1month, 2 months, 3 months, and 6 months.
  Scores from EQ-5D 5L questionnaire is assessed and compared.
Mean change in VisQoL scores | Baseline, 1 day, 1 week, 1month, 2 months, 3 months, and 6 months.
  Scores from VisQoL questionnaire is assessed and compared.
Mean change in wavefront aberrations | Baseline, 1 day, 1 week, 1month, 2 months, 3 months, and 6 months.
  Mean deviation (MD) of wavefront aberrations is assessed by Nidek OPD Scan III and compared.
Mean change in ocular surface and tear-film | Baseline, 1 day, 1 week, 1month, 2 months, 3 months, and 6 months.
  Mean deviation (MD) of ocular surface and tear-film parameters is assessed by Oculus Keratographer test and compared.
Mean change in vessel density | Baseline, 1 day, 1 week, 1month, 2 months, 3 months, and 6 months.
  Mean deviation (MD) of vessel density is assessed by Spectralis OCT2, Heidelberg-Engineering test and compared.
Side effects | Baseline, 1 day, 1 week, 1month, 2 months, 3 months, and 6 months.
  Side effects are measured by a review of the participant's medical and ophthalmic history.
People meeting driving standards | Baseline, 1 day, 1 week, 1month, 2 months, 3 months, and 6 months.
  Percentage (%) of people meeting driving standards is assessed by an Esterman binocular visual field test and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Wei He, Study Chair — He Eye Specialist Hospital, Shenyang.; Jun Li, Principal Investigator — He Eye Specialist Hospital, Shenyang.; Emmanuel E Pazo, Study Director — He Eye Specialist Hospital, Shenyang.
Locations (1):
- He Eye Specialist Hospital, Shenyang, Liaoning, China